CLINICAL TRIAL: NCT00476892
Title: A Multi-centre Randomised Controlled Trial of a Pelvic Floor Muscle Training Intervention for Women With Pelvic Organ Prolapse
Brief Title: Multi-centre Randomised Controlled Trial of Pelvic Floor Muscle Training for Prolapse
Acronym: POPPY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Glasgow Caledonian University (Other)
Collaborators: Chief Scientist Office of the Scottish Government (Other Government); South Glasgow University Hospitals NHS Trust (Other); University of Aberdeen (Other); University of Otago (Other)
Responsible Party: Dr Suzanne Hagen, NMAHP Research Unit, Glasgow Caledonian University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CZH/4/377; ISRCTN35911035
Record Dates: First submitted 2007-05-18; First posted 2007-05-22 (Estimated); Last update posted 2011-03-23 (Estimated); Status verified 2010-02

CONDITIONS: Pelvic Organ Prolapse
Keywords: Pelvic organ prolapse; Pelvic floor muscle training; Prolapse symptoms; Urinary symptoms; Sexual function; randomised controlled trial
MeSH Terms: conditions — Pelvic Organ Prolapse

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Other): It consists of five outpatient appointments (weeks 0, 2, 6, 11 and 16) with a local trial physiotherapist at a trial centre. At the first appointment a standardised history is taken from the woman, anatomy and function of the pelvic floor muscles are taught, and types of prolapse described, using diagrams and a model pelvis. Women are taught how to contract the muscles, and also how to contract and hold prior to an event that increases intra-abdominal pressure ("the Knack"). Pelvic floor muscles are assessed by vaginal examination and recorded on a dedicated form at each appointment thus determining the content of a single set of exercises for each woman. At least three sets of exercises daily is recommended. Women use an exercise diary to record compliance. Tailored advice is given on ways of reducing intra-abdominal pressure, e.g. advice on weight loss, chronic cough, heavy lifting and general exercise.
  Interventions: Procedure: Pelvic Floor Muscle Training
- 2 (No Intervention): Women allocated to the control group will be sent a lifestyle advice leaflet only, and will have no planned contact with the centre until their consultant review appointment at six months. The leaflet gives instructions on seeking advice where appropriate about weight loss, constipation, and avoidance of heavy lifting, coughing and high impact exercise, with a view to minimising increases in intra-abdominal pressure which may cause prolapse to worsen.

INTERVENTIONS:
Procedure: Pelvic Floor Muscle Training — Women in the intervention group attend 5 physiotherapy sessions. At each appointment a clinical history is taken, pelvic floor muscle assessment carried out, exercises taught and prescribed, and appropriate lifestyle advice given. At the first of these appointments a detailed explanation of the pelvic anatomy and different types of prolapse is given.
  Arms: 1

SUMMARY:
The aim of this study is to determine the effectiveness and cost-effectiveness of pelvic floor muscle training in the management of pelvic organ prolapse in women.

DETAILED DESCRIPTION:
Pelvic organ prolapse is a common problem that adversely affects the daily activities and quality of life of many women. Pelvic floor muscle training interventions are commonly used by physiotherapists to manage prolapse. However, a Cochrane review found limited evidence to support the effectiveness of such interventions. Based on the findings of a successful feasibility study, this multi-centre randomised controlled trial will address the paucity of evidence. 556 symptomatic women with diagnosed prolapse will be enrolled in 16 UK centres and 1 New Zealand centre over 16 months and randomised to pelvic floor muscle training plus lifestyle advice, or to receive a lifestyle leaflet only. Principal measures of outcome are: prolapse symptoms, prolapse severity, and subsequent further treatment up to 12 months after trial entry.

ELIGIBILITY:
Inclusion Criteria:

* New attendee at outpatient gynaecology clinic
* Any type of prolapse

Exclusion Criteria:

* Stage 0 or IV prolapse
* Women reporting no symptoms of prolapse
* Previous treatment for prolapse (surgery or formal instruction in Pelvic Floor Muscle Training [PMFT,]unless completed more than 5 years ago, pessary, unless pessary removed more than 12 months ago)
* Unable to comply with PFMT
* women who have urogenital atrophy requiring treatment with local oestrogens (after an 8 week course of local oestrogen such women can be included);
* Pregnant or less than 6 months post-natal
* Unable to give informed consent

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 448 (Actual)
Dates: Start 2007-06; Primary Completion 2010-07 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Prolapse symptom score (questions developed in feasibility study and undergoing validation). Primary economic outcome measures are: use of health services, average number of days of prolapse symptoms and further prolapse treatment needed/received | 1 year

SECONDARY OUTCOMES:
Prolapse-related quality of life, prolapse severity, need for further prolapse treatment. Other outcomes include: lifestyle changes, urinary symptoms, bowel symptoms, sexual symptoms, general health status. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Suzanne Hagen, Principal Investigator — NMAHP Research Unit, Glasgow Caledonian University
Locations (28):
- St George Hospital, Sydney, Australia
- Ireland (2):
  - Antrim Area Hospital, Antrim
  - Belfast City Hospital, Belfast
- Dunedin School of Medicine, Dunedin, New Zealand
- United Kingdom (24):
  - Crosshouse Hospital / Ayrshire Maternity Hospital, Kilmarnock, Ayrshire
  - Forth Park Hospital, Kirkcaldy, Fife
  - Aberdeen Royal Infirmary, Aberdeen, Grampian
  - North Hampshire Hospitals NHS Trust, Basingstoke, Hampshire
  - Royal Infirmary of Edinburgh, Edinburgh, Lothian
  - St John's Hospital, Livingston, West Lothian
  - Birmingham Women's Hospital, Birmingham
  - Bradford Royal Infirmary, Bradford
  - Addenbrooke's Hospital, Cambridge
  - Chester Hospital, Chester
  - St Richard's Hospital, Chichester
  - Ninewells Hospital, Dundee
  - Falkirk and District Royal Infirmary, Falkirk
  - Western Infirmary, Glasgow
  - Glasgow Royal Infirmary, Glasgow
  - Victoria Infirmary, Glasgow
  - Southern General Hospital, Glasgow
  - Castle Hill Hospital, Hull
  - St James's University Hospital, Leeds
  - St Mary's Hospital, Manchester
  - Borders General Hospital, Melrose
  - James Cook University Hospital, Middlesbrough
  - Worcestershire Royal Hospital, Worcester
  - York Hospital, York